CLINICAL TRIAL: NCT04028700
Title: Red Blood Cell Survival Study: The Impact of Oxidative Stress on Erythrocyte Biology
Brief Title: The Impact of Oxidative Stress on Erythrocyte Biology
Acronym: RBC Survival
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding not renewed
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Columbia University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-0587; R01HL148151-01 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease Without Crisis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will not be told which type of blood they are receiving first. There is no way to tell if blood has enzyme deficiencies by looking at it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- G6PD Deficient Red Blood Cell Transfusion, then Non-G6PD deficient Red Blood Cell Transfusion (Experimental): Transfusion of a red blood cell unit that has been identified by local laboratory procedures to be deficient in G6PD enzyme activity followed after 4 months by transfusion of a red blood cell unit that has been identified by local laboratory procedures to not be deficient in G6PD enzyme activity.
  Interventions: Biological: G6PD Deficient Red Blood Cell Transfusion; Biological: Non-G6PD deficient Red Blood Cell Transfusion
- Non-G6PD deficient Red Blood Cell Transfusion, then G6PD Deficient Red Blood Cell Transfusion, (Active Comparator): Transfusion of a red blood cell unit that has been identified by local laboratory procedures to not be deficient in G6PD enzyme activity followed after 4 months by transfusion of a red blood cell unit that has been identified by local laboratory procedures to be deficient in G6PD enzyme activity
  Interventions: Biological: G6PD Deficient Red Blood Cell Transfusion; Biological: Non-G6PD deficient Red Blood Cell Transfusion

INTERVENTIONS:
Biological: G6PD Deficient Red Blood Cell Transfusion — Patients will receive a red blood cell transfusion. The last 50 mL of the transfusion will be labeled with chromium to allow investigators to study the lifespan of the red blood cells transfused into each patient.
Biological: Non-G6PD deficient Red Blood Cell Transfusion — Patients will receive a red blood cell transfusion. The last 50 mL of the transfusion will be labeled with chromium to allow investigators to study the lifespan of the red blood cells transfused into each patient.

SUMMARY:
This study will address if red blood cells transfused to a sickle cell patient from a donor with a glucose-6-phosphate-dehydrogenase (G6PD) enzyme deficiency have a different lifespan as measured by the percentage of red blood cells that survive post-transfusion compared to red blood cells transfused to a sickle cell patient from a donor without a G6PD enzyme deficiency.

DETAILED DESCRIPTION:
This prospective, phase II, crossover, single-blind, randomized transfusion order study will address if red blood cells from donors with a G6PD enzyme deficiency have a different lifespan once transfused into a patient with sickle cell disease than red blood cells from an otherwise normal donor. Results of this critical study will guide future research and donor testing policies to ensure that patients receive the most appropriate units of blood for their condition. Each patient randomized to the study will receive 2 blood transfusions, one from a G6PD deficient donor and one from an otherwise normal donor. Half the patients (8) will receive G6PD deficient blood first while the other half (8) will receive non-G6PD deficient blood first. Patients will have a wash-out period of at least 4 months before receiving the opposite type of blood transfusion. The blood transfusion order will be randomized. There is currently no standard of testing in place to screen blood donations for G6PD enzyme deficiency. It is believed that up to 10% of the antigen-matched donors for patients with sickle cell disease are G6PD deficient, and the lifespan is unknown in the sickle cell population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Has diagnosis of sickle cell disease
* Steady state (no pain or baseline pain and ≥1 month from any hospital admission)
* Receiving chronic transfusions (i.e., regular transfusion every 4-8 weeks).

Exclusion Criteria:

* History of transfusion reactions not adequately managed by antihistamines
* Does not have crossmatch compatible red cells
* Known G6PD deficiency
* Hepato- or splenomegaly
* Participation in another therapeutic trial
* Pregnant or nursing
* HIV positive
* At investigator discretion for uncontrolled inter-current illness or social situation limiting compliance with study requirements.
* Inability to speak and/or read English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Karafin, MD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator proposing to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- G6PD Deficient Red Blood Cell Transfusion, Then Non-G6PD Deficient Red Blood Cell Transfusion: Transfusion of a red blood cell unit that has been identified by local laboratory procedures to be deficient in glucose-6-phosphate-dehydrogenase (G6PD) enzyme activity followed after 4 months by transfusion of a red blood cell unit that has been identified by local laboratory procedures to not be deficient in G6PD enzyme activity.
  G6PD Deficient Red Blood Cell Transfusion: Patients will receive a red blood cell transfusion. The last 50 mL of the transfusion will be labeled with chromium to allow investigators to study the lifespan of the red blood cells transfused into each patient.
  Non-G6PD deficient Red Blood Cell Transfusion: Patients will receive a red blood cell transfusion. The last 50 mL of the transfusion will be labeled with chromium to allow investigators to study the lifespan of the red blood cells transfused into each patient.
Period: Initial Intervention
Arm/Group | G6PD Deficient Red Blood Cell Transfusion, Then Non-G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion, Then G6PD Deficient Red Blood Cell Transfusion,
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Washout (4 Months)
Arm/Group | G6PD Deficient Red Blood Cell Transfusion, Then Non-G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion, Then G6PD Deficient Red Blood Cell Transfusion,
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | G6PD Deficient Red Blood Cell Transfusion, Then Non-G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion, Then G6PD Deficient Red Blood Cell Transfusion,
Started (Study was teminated before the Second Intervention began.) | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G6PD Deficient Red Blood Cell Transfusion, Then Non-G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion, Then G6PD Deficient Red Blood Cell Transfusion, | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Red Blood Cells Surviving
Description: Post-Transfusion Recovery
Time Frame: 24 hours post-transfusion
Measure: Mean (Standard Deviation); unit: percentage of surviving red cells
Groups:
- G6PD Deficient Red Blood Cell Transfusion: Transfusion of a red blood cell unit that has been identified by local laboratory procedures to be deficient in G6PD enzyme activity.
  G6PD Deficient Red Blood Cell Transfusion: Patients will receive a red blood cell transfusion. The last 50 mL of the transfusion will be labeled with chromium to allow investigators to study the lifespan of the red blood cells transfused into each patient.
- Non-G6PD Deficient Red Blood Cell Transfusion: Transfusion of a red blood cell unit that has been identified by local laboratory procedures to not be deficient in G6PD enzyme activity.
  Non-G6PD deficient Red Blood Cell Transfusion: Patients will receive a red blood cell transfusion. The last 50 mL of the transfusion will be labeled with chromium to allow investigators to study the lifespan of the red blood cells transfused into each patient.
Arm/Group | G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion
Number analyzed (Participants) | 3 | 5
percentage of surviving red cells | 82.91 (5.57) | 91.03 (3.90)

2. Secondary Outcome: Mean Percent Change in Hemoglobin A
Description: Hemoglobin A
Time Frame: 1 hour post-transfusion, 4 weeks post-transfusion
Measure: Mean (Standard Deviation); unit: Percentage of Hemoglobin A
Arm/Group | G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion
Number analyzed (Participants) | 3 | 5
Percentage of Hemoglobin A | 25.87 (8.14) | 21.02 (3.55)

ADVERSE EVENTS:
Time Frame: From the time of chromium infusion until the end the last blood draw, a total of approximately 4 weeks.
Arm/Group | G6PD Deficient Red Blood Cell Transfusion | Non-G6PD Deficient Red Blood Cell Transfusion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G6PD Deficient Red Blood Cell Transfusion (N=3) | Non-G6PD Deficient Red Blood Cell Transfusion (N=5)
Shortness of Breath due to Heart Palpitations (Cardiac disorders) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stuffy Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Headache (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04028700/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04028700/ICF_000.pdf